CLINICAL TRIAL: NCT00691158
Title: A Pilot Study of the fMRI Response to Leptin and Pramlintide
Brief Title: A Study of the Functional Magnetic Resonance Imaging Response to Leptin and Pramlintide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan Purnell, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: eIRB #2168; OCTRI #933 (Other: Oregon Health and Sciences University)
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — pramlintide; Islet Amyloid Polypeptide; Saline Solution; Leptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1- Normal Saline (Placebo Comparator): 4.7 mls normal saline IV bolus
  Interventions: Drug: Placebo (Normal Saline)
- 2 Metreleptin (Active Comparator): IV Leptin bolus
  Interventions: Drug: 2 Metreleptin
- 3 Pramlintide (Active Comparator): IV Pramlintide bolus at Timpoint +0 and +30 minutes
  Interventions: Drug: Pramlintide (Amylin)
- 4 Leptin plus Pramlintide (Active Comparator): leptin and pramlintide IV bolus injection at timpoints 0 and +30 minutes
  Interventions: Drug: Leptin plus Pramlintide

INTERVENTIONS:
Drug: Pramlintide (Amylin) — 4.7 mls of Amylin 15mcg/ml IV bolus.
  Other Names: Amylin
  Arms: 3 Pramlintide
Drug: Placebo (Normal Saline) — 4.7 mls normal saline IV bolus x1
  Other Names: Placebo
  Arms: 1- Normal Saline
Drug: 2 Metreleptin — Receive .06mg/kg of metreleptin IV bolus x1
  Other Names: Leptin
  Arms: 2 Metreleptin
Drug: Leptin plus Pramlintide — receive leptin IV bolus x1 and pramlintide bolus at Timepoint +0 and +30 minutes.
  Other Names: Leptin and Amylin
  Arms: 4 Leptin plus Pramlintide

SUMMARY:
The purpose of this study is to identify how certain parts of the brain that help control body weight respond to an infusion of hormones called leptin and amylin.

DETAILED DESCRIPTION:
Following an overnight fast, subjects will undergo fMRI measurements of the hypothalamus, brainstem and whole brain during an infusion of either normal saline, pramlintide, leptin, or the combination leptin and pramlintide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year to 45 years of age
* MI 18 to 25 kg/m2 or ≥ 30 kg/m2
* At maximal lifetime weight
* Weight stable for at least 3 months

Exclusion Criteria:

* Those with a major medical illness or who require prescription medication, including: cancer, coronary artery disease, hypertension, and diabetes.
* Subjects taking psychiatric or centrally-acting (CNS) medications or who are diagnosed with a psychiatric or neurological illness, including:

  * depression
  * anorexia
  * bulimia
  * seizure disorder.
* Exercise > 30 minutes, 3 times a week
* Alcohol consumption > 2 drinks / day
* Weight > 350 lbs (159 kg) (weight limit for MR machine)
* Illicit drug use
* Pregnancy
* Extreme dietary habits as determined by a GCRC nutritionist: very high or low dietary carbohydrate or fat intakes
* Those with a contraindication to exposure to strong magnetic fields: presence of metal in the body such as body piercing, shrapnel, cardiac pacemakers or aneurysm clips
* Those with claustrophobia
* Anaphylaxis and known hypersensitivity to E. coli-derived proteins
* Allergies or contraindications to metreleptin or pramlintide
* Renal or hepatic impairment
* Women who are lactating
* Tobacco use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-01; Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
To measure the fMRI response in the hypothalamus and brainstem, and whole brain, to intravenous leptin, pramlintide, combination leptin and pramlintide, and saline control. | over 90 minutes
  measurements at each study time are include fMRI, blood draws and Visual Analog Score.

SECONDARY OUTCOMES:
Timed blood samples during infusion will establish the time course for peak levels of infused hormones as well as detectable changes in insulin and glucose levels. | over 90 minutes
  Blood samples are taken every 5 minutes from Timepoint +0 to Timepoint +60 and again one time at Timepoint +90

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, M.D., Principal Investigator — OHSU - Center for the Study of Weight Regulation
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States